CLINICAL TRIAL: NCT04272099
Title: Individual and Social Determinants of Health in Global Pediatric Diabetes Care Delivery - a Participatory Search for Barriers and Opportunities
Brief Title: Social Determinants of Global Pediatric Diabetes
Acronym: DESIDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, julia.vonoettingen, Assistant Professor at McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2018-3350
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus
Keywords: Adolescent; Child; Quality of Life; Self Efficacy; Haiti; Emigrants and Immigrants; Canada
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PG1 (patients with diabetes 0-25 years of age): Patients 0 to 25 years of age, with a diagnosis of diabetes that are either followed at Kay Mackenson Pediatric Clinic, Haiti, or who are of Haitian ancestry, defined as both maternal and paternal grandparents being born in Haiti, and attend one of the three diabetes clinics in Montreal.
  Interventions: Other: Administration of standardized questionnaires; Device: Physical activity tracker; Other: Dietary log
- PG2 (patient's principal caregiver): The patient's principal caregiver (a parent of legal guardian).
  Interventions: Other: Administration of standardized questionnaires

INTERVENTIONS:
Other: Administration of standardized questionnaires — Administration of questionnaires assessing subjective socioeconomic status (SES), health literacy, perceived health, health related quality of life, self-esteem and diabetes self-efficacy
Device: Physical activity tracker — PG1 will be asked to wear a physical activity tracker for one week to monitor activity patterns including walking distance, calorie expenditure, sedentary time and sleep.
  Groups: PG1 (patients with diabetes 0-25 years of age)
Other: Dietary log — PG1 (or PG2 as proxies when appropriate) will report to a study coordinator via phone a full dietary log of PG1 once per week on rotating days of the week for three weeks.
  Groups: PG1 (patients with diabetes 0-25 years of age)

SUMMARY:
There is little data from low-income countries on setting and culture specific perception of childhood diabetes and disease specific stressors including stigma, and how these may affect disease related quality of life, coping strategies, self-efficacy and glycemic control.

The goal of this study is to understand how socioeconomic, psychosocial, cultural, and diet and activity related factors in children and adolescents with diabetes in Haiti relate to quality of life, self-efficacy and glycemic control, and comparing the factor analysis to immigrant children of Haitian ancestry with diabetes living in Montreal.

An innovative, participatory research approach will allow for a holistic evaluation of modifiable barriers to optimal pediatric diabetes care delivery in resource limited settings, while providing translational information for care delivery of diabetes in underserved, immigrant populations in high-income settings.

DETAILED DESCRIPTION:
Pediatric diabetes is a lifelong condition that affects an estimated 542,000 children under the age of 14 years worldwide, of whom the majority live in low- and middle-income countries. Epidemiological data from Haiti on the incidence and prevalence of diabetes in childhood are currently being collected. In Haiti, as in many other low-income countries, there is likely to be incomplete case ascertainment due to a lack of accurate and timely diagnosis. The investigators' group as well as others have observed remarkable differences in clinical presentation of childhood diabetes as compared to Caucasian patients. Presentations reminiscent of "atypical" diabetes, fibrocalculous pancreatitis, and malnutrition related diabetes seem to be more frequent. Many patients retain low exogenous insulin requirements past 5-10 years after initial diagnosis, suggesting much longer periods of residual endogenous insulin production as compared to Caucasian patients. Further, while complications of diabetes are considered a rarity in Caucasian patients, up to 20% of Haitian children and adolescents presenting with diabetes have eye complications (cataract and/or retinopathy) at the time of or within 2-3 years of diagnosis (unpublished data). Although genetic, environmental and immune factors have been hypothesized, the investigators do not currently understand the underlying etiology of these unusual phenotypes, and how those relate to glycemic control.

Limited data from sites in low-income countries where pediatric diabetes care has been established (including from Haiti) concerningly show that even when patients are regularly followed and insulin and diabetes care supplies are provided free of charge, glycemic control remains suboptimal. While psychosocial, sociocultural, educational and economic factors (including diet habits and food insecurity) are known to be associated with glycemic control, detailed evaluations from low-income countries on these factors and how they related to diabetes management in children are lacking. Similarly, there is little data from low-income countries on setting and culture specific perception of childhood diabetes and disease specific stressors including stigma, and how these may affect disease related quality of life, coping strategies, self-efficacy and glycemic control.

Child and parent health literacy, defined as "the degree to which individuals have the capacity to obtain, process, and understand basic health information and services needed to make appropriate health decisions" has been shown to impact diabetes self-efficacy, including improved diabetes management and glycemic control. However, little is known about health literacy in children with diabetes and their families in resource limited settings, and its effect on diabetes care has not been evaluated in Haiti. The degree to which these complex, interrelated and dynamic factors affect long-term outcomes is not known.

Lastly, community, family and peer support is known to impact health outcomes in children with chronic disease. However, in many resource limited settings local support groups are not available, or are only offered at the diabetes clinic, which can be remote from the patient's home (many patients travel several hours to get to the diabetes clinic). It is unknown if the use of social networks for patients with diabetes in resource limited settings can improve perceived and objective health related outcomes.

The specific aims of this research project are:

1. To evaluate the socioeconomic status (SES) of children with diabetes and their families in Haiti, and of Haitian immigrant children with diabetes in Montreal.
2. To conduct a detailed psychosocial evaluation of participating children.
3. To analyze macro- and micronutrient intake, dietary patterns, food security and physical activity patterns in participating children.
4. To investigate perceptions and explanations of illness and health, and to assess health literacy and diabetes self-efficacy in participating children and caregivers.
5. To evaluate how SES, psychosocial well-being, illness perception, health literally, self-efficacy and lifestyle habits relate to glycemic control and quality of life and clinical phenotypes.

The investigators will also assess how results compare between the two study sites.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for PG1 are age 0-25 years, be of Haitian ancestry defined as having both maternal and paternal grandparents being born in Haiti, have a diagnosis of diabetes, and are enrolled in one of the two study site clinics.
* Inclusion criteria for PG2 are being the principal caregiver for a PG1.

Exclusion Criteria:

* Exclusion criteria for PG1 and PG2 are inability to provide informed consent (if 18 years or older) or inability of a parent or legal guardian to provide informed consent (if younger than 18 years).

Ages: 0 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will take place at 2 sites:
  * Haiti, through the Kay Mackenson Clinic (KMC) in Montrouis (with a catchment area across the country),
  * Montreal, through the diabetes clinics of the Montreal Children's Hospital (MCH), the CHU Sainte-Justine Hospital (CHUSJ) and the Centre intégré universitaire de santé et de services sociaux de l'Est-de-l'Île-de-Montréal (CIUSSS) in Montreal, Canada. Participants will be enrolled from each local clinic.
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Socioeconomic status, health literacy level, and diabetes self-efficacy in PG1 and PG2 | These variables will be assessed cross-sectionally at time of enrolment
  ZIP code-based SES indicators and questionnaires on health literacy, and diabetes self-efficacy
The psychosocial and physical health status of PG1 | These variables will be assessed cross-sectionally at time of enrolment
  Questionnaires on perceived health, health-related quality of life, and self-esteem
Diet and activity related lifestyle habits of children with diabetes of PG1 | These variables will be assessed prospectively over three months during follow-up from time of enrolment
  Collection of data on dietary composition, meal distribution pattern, and activity patterns including walking distance, calorie expenditure, sedentary time and sleep.
Glycemic control, health related quality of life and clinical phenotypes of PG1 | Retrospective data from time of diagnosis, cross-sectional at time of enrolment and prospective monitoring over three months from time of diabetes diagnosis and over three months from time of enrolment
  Extraction of clinical records, data on the date of diagnosis, clinical presentation at diagnosis, hemoglobin A1C measurements over time, most recent weight, height, body mass index (BMI) and total daily insulin dose. Questionnaire on health-related quality of life. Data collection on blood glucose monitoring frequency and distribution, blood glucose values, as well as insulin dosing and injections.

SECONDARY OUTCOMES:
Psychometric evaluation of the health literacy, health-related quality of life, self-esteem and self-efficacy questionnaires in PG1 | Cross-sectional assessment at time of enrolment
  Standardized questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Julia von Oettingen, MD PhD MMSc, Principal Investigator — MUHC-RIMUCH
Locations (4):
- Canada (3):
  - Centre intégré universitaire de santé et de services sociaux de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
- Kay Mackenson Pediatric Clinic, Montrouis, Artibonite, Haiti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall SL, Edidin D, Sharma V, Ogle G, Arena VC, Orchard T. Current clinical status, glucose control, and complication rates of children and youth with type 1 diabetes in Rwanda. Pediatr Diabetes. 2013 May;14(3):217-26. doi: 10.1111/pedi.12007. Epub 2012 Dec 28. PMID 23279222
- [Background] Marshall SL, Edidin DV, Arena VC, Becker DJ, Bunker CH, Gishoma C, Gishoma F, LaPorte RE, Kaberuka V, Ogle G, Sibomana L, Orchard TJ. Glucose control in Rwandan youth with type 1 diabetes following establishment of systematic, HbA1c based, care and education. Diabetes Res Clin Pract. 2015 Jan;107(1):113-22. doi: 10.1016/j.diabres.2014.09.045. Epub 2014 Oct 7. PMID 25458328
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Piloya-Were T, Sunni M, Ogle GD, Moran A. Childhood diabetes in Africa. Curr Opin Endocrinol Diabetes Obes. 2016 Aug;23(4):306-11. doi: 10.1097/MED.0000000000000262. PMID 27228228
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Goodman E, Adler NE, Kawachi I, Frazier AL, Huang B, Colditz GA. Adolescents' perceptions of social status: development and evaluation of a new indicator. Pediatrics. 2001 Aug;108(2):E31. doi: 10.1542/peds.108.2.e31. PMID 11483841
- See also: International Diabetes Federation. IDF World Diabetes Atlas 2015 — http://www.diabetesatlas.org